CLINICAL TRIAL: NCT05365659
Title: A Phase 1 Cohort Dose Escalation and Expansion Trial to Determine the Safety, Tolerance, Maximum Tolerated Dose, and Preliminary Antineoplastic Activity of IKS03 in Patients With Advanced B Cell Non-Hodgkin Lymphomas (NHL)
Brief Title: IKS03 in Patients With Advanced B Cell Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Iksuda Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IKS03-01
Record Dates: First submitted 2022-05-02; First posted 2022-05-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: B-cell Non-Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; B-cell Lymphoma
Keywords: CD19; non-Hodgkin lymphoma; NHL; DLBCL; MCL; advance lymphoma; IKS03; lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose Escalation Cohort (Part 1) (Experimental): Each patient will receive repeat doses (by intravenous (IV) infusions) on Day 1 of each 21-day cycle. Participants may continue on study until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: IKS03
- Dose Expansion: Diffuse-Large B-Cell Lymphoma Participants (Experimental): Each patient will receive IKS03 at the recommended dose for expansion (RDE) defined in Part 1 on Day 1 of each 21-day cycle. Participants may continue on study until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: IKS03
- Dose Expansion: Follicular Cell Lymphoma Participants (Experimental): Each patient will receive IKS03 at the recommended dose for expansion (RDE) defined in Part 1 on Day 1 of each 21-day cycle. Participants may continue on study until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: IKS03
- Dose Expansion: Mantle Cell Lymphoma Participants (Experimental): Each patient will receive IKS03 at the recommended dose for expansion (RDE) defined in Part 1 on Day 1 of each 21-day cycle. Participants may continue on study until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: IKS03
- Dose Expansion: Other B cell lymphoma (B-NHL not otherwise specified [NOS]) (Experimental): Each patient will receive IKS03 at the recommended dose for expansion (RDE) defined in Part 1 on Day 1 of each 21-day cycle. Participants may continue on study until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: IKS03

INTERVENTIONS:
Drug: IKS03 — IKS03 is a human monoclonal antibody (Ab) targeting CD19 linked to a pyrrolobenzodiazepine (PBD) pro-drug as the cytotoxic agent.

SUMMARY:
This first-in-human study will evaluate the recommended dose for further clinical development, safety, tolerability, antineoplastic activity, immunogenicity, pharmacokinetics and pharmacodynamics of IKS03, a CD19 targeting antibody-drug conjugate, in patients with advanced B cell non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
The study will consist of 2 parts: dose-escalation (Part 1) and dose-expansion (Part 2). The dose-escalation part (Part 1) of the study is to evaluate the safety and tolerability of increasing dose levels of IKS03 to establish a recommended dose for expansion (RDE); and the dose-expansion part (Part 2) of the study is to further evaluate the safety, pharmacokinetics/pharmacodynamics, and efficacy of IKS03 at the RDE.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 18 years of age
2. Part 1: documented B cell NHL (any subtype except Burkitt lymphoma, Waldenström macroglobulinemia, chronic lymphocytic leukemia); previously confirmed CD19-positive if feasible
3. Part 2: documented B cell NHL (subtypes to be determined); confirmed CD19-positive; possible expansion cohorts may include:

   1. Diffuse large B cell lymphoma (including germinal center B cell type, activated B cell type)
   2. Follicular lymphoma (including duodenal-type follicular lymphoma)
   3. Mantle cell lymphoma
   4. B cell lymphomas not specified
4. If B cell NHL subtype likely to have bone marrow involvement must be willing to undergo bone marrow biopsy in the event of an on-study complete response to confirm response
5. NHL that is relapsed, refractory to, or intolerant of existing therapy(ies) with known curative potential, or for which no standard therapy is available; must have received at least 2 prior lines of systemic therapy
6. Must be in need of systemic treatment and not require immediate cytoreductive therapy
7. Part 1: measurable or non-measurable disease
8. Part 2: measurable disease according to The Revised Criteria/Lugano Classification
9. Part 1: screening tumor biopsy requested, but optional; Part 2: patient must agree to screening tumor biopsy
10. ECOG performance status 0 or 1; anticipated life expectancy ≥ 10 weeks
11. Women of childbearing potential and fertile men agreeing to use two effective methods of contraception (including a highly effective method of contraception); women beginning 2 weeks prior to the first dose, men beginning prior to the first dose, and both continuing until 8 months after the last dose of study drug; male patients must also agree to refrain from sperm donation during this period.
12. Ability to understand and give written informed consent

Exclusion Criteria:

1. Women who are pregnant or intending to become pregnant before, during, or within 8 months after the last dose of study drug; women who are breastfeeding
2. Patients documented to be CD19-negative
3. Central nervous system (CNS) lymphoma, leptomeningeal infiltration, or spinal cord compression not controlled by prior surgery or radiotherapy; symptoms suggesting CNS involvement
4. Part 2: History of another malignancy within 2 years, with the exception of:

   1. Treated, non-melanoma skin cancers
   2. Treated carcinoma in situ (e.g., breast, cervix)
   3. Controlled, superficial carcinoma of the urinary bladder
   4. T1a or b prostate carcinoma treated according to standard of care, with PSA within normal limits
   5. Papillary thyroid carcinoma Stage I treated surgically for cure
5. Any of the following hematologic abnormalities at baseline (transfusion allowed > 5 days previous):

   1. Hemoglobin < 8.0 g/dL
   2. Absolute neutrophil count < 1,000 per mm3
   3. Platelet count < 75,000 per mm3
6. Any of the following laboratory abnormalities at baseline:

   1. Total bilirubin > 1.5 × upper limit of normal (ULN); > 3 × ULN if with Gilbert's Syndrome
   2. AST or ALT > 3 × ULN; > 5 × ULN if due to hepatic involvement by tumor
   3. Estimated GFR ≤ 60 mL/min corrected for BSA
   4. Albuminuria defined as urine albumin to creatinine ratio < 30 mg/g or < 3 mg/mmol) by spot urine albumin
7. Any of the following coagulation parameter abnormalities at baseline unless on a stable dose of anticoagulant therapy for a prior thrombotic event:

   1. PT or INR > 1.5 × ULN; > 3× ULN if anticoagulated)
   2. PTT > 1.5 × ULN; > 3× ULN if anticoagulated
8. Any of the following laboratory abnormalities at baseline aimed at assessing renal function:

   1. Estimated glomerular filtration rate (eGFR) ≤ 60 mL/min, corrected for BSA.
   2. Albuminuria defined as urine albumin to creatinine ratio (UACR) ≥ 30 mg/g or ≥ 3 mg/mmol by spot urine albumin
9. Patients with:

   1. Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks unless adequately treated and stable
   2. Active uncontrolled bleeding or a known bleeding diathesis
10. Significant cardiovascular disease or condition, including:

    1. Congestive heart failure or angina pectoris requiring therapy
    2. Ventricular arrhythmia requiring therapy or other uncontrolled arrhythmia
    3. Severe conduction disturbance (e.g., 3rd degree heart block)
    4. QTc interval ≥ 480 milliseconds
    5. Left ventricular ejection fraction below the lower limit of normal or < 50% by MUGA scan or echocardiogram
    6. Class III or IV cardiovascular disease according to the New York Heart Association Functional Classification
    7. History of acute coronary syndromes (e.g., MI, unstable angina), coronary angioplasty, stenting, or bypass within 6 months
11. Significant liver disease, including:

    1. Non-infectious hepatitis
    2. Hepatic cirrhosis (Child-Pugh Class B and Class C)
12. Significant pulmonary disease or condition, including:

    1. Significant symptomatic COPD, as assessed by the Investigator
    2. History or any current evidence on imaging studies of interstitial lung disease, pulmonary fibrosis
    3. History of pulmonary inflammatory disease, pneumonitis, ARDS
    4. History of pneumonia within 6 months
13. Significant corneal disease or condition, including history of or current evidence of keratitis
14. Clinically significant CNS disease or condition including PML, epilepsy, vasculitis, or neurodegenerative disease. Also including TIA or stroke within 6 months
15. Known HIV infection or AIDS
16. Active hepatitis B virus or hepatitis C virus infection
17. Any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 2 weeks
18. Autoimmune disease or condition requiring systemic steroids or other immunosuppressive medications
19. Unresolved Grade > 1 AE associated with any prior antineoplastic therapy (except persistent Grade 2 alopecia, peripheral neuropathy, decreased hemoglobin, neutropenia, lymphopenia, hypomagnesemia, and/or endocrine end-organ failure being adequately managed by HRT)
20. Known or suspected hypersensitivity to any of the excipients of formulated study drug
21. Inadequate recovery from a surgical procedure, or a major surgical procedure within 4 weeks
22. Any other serious, life-threatening, or unstable preexisting medical condition, including significant organ system dysfunction, or clinically significant laboratory abnormality(ies)
23. A psychiatric disorder or altered mental status that would preclude understanding of the informed consent process

Drugs and Other Treatments to be Excluded:

1. Receipt of:

   1. Any CD19-targeted therapy within 3 months
   2. Any tumor vaccine within 6 weeks (must have progressed if previously received)
2. Prior autologous/allogeneic CAR-T therapy if known to be CD19-negative after
3. Any other antineoplastic agent for the primary malignancy without delayed toxicity within 4 weeks or 5 plasma half-lives, whichever is shortest (except nitrosoureas and mitomycin C within 6 weeks)
4. Any other investigational treatments within 4 weeks
5. Drugs known to impair renal function, including:

   1. NSAIDS within 3 days
   2. Aminoglycoside antibiotics, amphotericin B, etc. within 1 week
   3. Bisphosphonates within 1 month
6. Prior solid organ transplant
7. Allogeneic HSCT within 6 months, or:

   1. If receiving immunosuppression
   2. If with active evidence of GVHD
8. Autologous hematopoietic stem cell transplantation (HSCT) within 3 months
9. Radiotherapy:

   1. To target lesions within 4 weeks unless progression of the lesion has been documented
   2. To non-target lesions within 1 week
10. Live/live-attenuated vaccines against infectious diseases within 4 weeks
11. Immunosuppressive or systemic glucocorticoid therapy (> 10 mg prednisone daily or equivalent) within 2 weeks
12. Prophylactic use of hematopoietic growth factors within 1 week
13. Herbal therapies and supplements within 2 weeks
14. Strong inhibitors of cytochrome P450 within 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Recommended Dose for Expansion (Part 1) | Up to 20 months
  RDE will be determined using dose limiting toxicities (DLTs) and all other available study data
Objective Response Rate (Part 2) | up to 42 months
  Antineoplastic effects will be assessed by Criteria for Response Assessment: The Lugano Classification (Cheson 2014)

SECONDARY OUTCOMES:
Evaluation of the immunogenicity of IKS03 (Part 1 and 2) | Up to 42 months
  Occurrence of ADA measured in serum at selected timepoints during the study
Plasma Concentrations of IKS03 (Part 1 and 2) | Up to 42 months
  Pharmacokinetic profile will be characterized by concentrations of IKS03
Determine recommended Phase 2 dose (RP2D) (Part 2) | Up to 42 months
  Based on evidence of antitumor activity, acceptable tolerability, evidence of achieving target plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Paul I Nadler, MD, Study Director — Iksuda Therapeutics
Locations (13):
- University of Maryland Baltimore, Baltimore, Maryland, United States
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Linear Clinical Research, Perth, Western Australia
- Jewish General Hospital, Montreal, Quebec, Canada
- Italy (4):
  - La Fondazione e l'Istituto di Candiolo, Candiolo
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) Ospedale San Raffaele, Milan
  - Istituto Europeo Clinico Humanitas, Milan
  - Istituto Europeo di Oncologia, Milan
- Spain (3):
  - Institut Catala D'Oncologia, Badalona
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No